CLINICAL TRIAL: NCT04965844
Title: Safety and Efficacy of a Closed-loop Oxygen Control for High Flow Nasal Therapy in ICU Patients: a Randomized Cross-over Study (The HILOOP Study)
Brief Title: Closed-loop Oxygen Control for High Flow Nasal Therapy
Acronym: HILOOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PR(AG)539/2020
Record Dates: First submitted 2021-05-04; First posted 2021-07-16 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-10

CONDITIONS: High Flow Nasal Cannula; Oxygen Therapy; Hypoxemia; Hyperoxemia; Acute Respiratory Failure; Respiratory Insufficiency
Keywords: High flow nasal cannula; Nasal high flow; Oxygen close-loop; Hypoxemia; Hyperoxemia
MeSH Terms: conditions — Hypoxia; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen close-loop (Experimental): Four hours period where the fraction of inspired oxygen delivered will be automatically titrated based on SpO2 values.
  Interventions: Device: Oxygen close-loop
- Manual FiO2 adjustment (Active Comparator): Four hours period where the fraction of inspired oxygen delivered will be manually adjusted by the healthcare personnel based on SpO2 values.
  Interventions: Device: No intervention

INTERVENTIONS:
Device: Oxygen close-loop — The Automatic FiO2 option provides automated adjustment of the ventilator Oxygen setting to maintain the patient's SpO2 in a defined target range. When using the software option, the user defines the SpO2 target range, as well as the SpO2 emergency limits, and the device adjusts the Oxygen setting to keep the patient's SpO2 in the target range.
  Arms: Oxygen close-loop
Device: No intervention — Manual FiO2 adjustment according to SpO2 values
  Arms: Manual FiO2 adjustment

SUMMARY:
In patients with acute hypoxemic respiratory failure (AHRF), High Flow Nasal Therapy (HFNT) improves oxygenation, tolerance, and decrease work of breathing as compared to standard oxygen therapy by facemask. Current guidelines recommend adjusting oxygen flow rates to keep the oxygen saturation measured by pulse oximetry (SpO2) in the target range and avoid hypoxemia and hyperoxemia. The hypothesis of the study is that closed loop oxygen control increases the time spent within clinically targeted SpO2 ranges and decreases the time spent outside clinical target SpO2 ranges as compared to manual oxygen control in ICU patients treated with HFNT.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>17yo) patients admitted to the ICU treated with HFNT for at least 8h
* Requiring FiO2 ≥ 30% to keep SpO2 in the target ranges defined by the clinician
* Written informed consent signed and dated by the patient or one relative in case that the patient is unable to consent, after full explanation of the study by the investigator and prior to study participation.

Exclusion Criteria:

* Patient with indication for immediate continuous positive airway pressure (CPAP), noninvasive ventilation (NIV), or invasive mechanical ventilation
* Hemodynamic instability defined as a need of continuous infusion of epinephrine or norepinephrine > 1 mg/h
* Low quality on the SpO2 measurement using finger and ear sensor (quality index below 60% on the Massimo SpO2 sensor, which is displayed by a red or orange colour bar)
* Severe acidosis (pH ≤ 7.30)
* Pregnant woman
* Patients deemed at high risk for need of mechanical ventilation within the next 8 hours
* Chronic or acute dyshemoglobinemia: methemoglobin, carbon monoxide (CO) poisoning, sickle cell disease
* Tracheotomised patient
* Formalized ethical decision to withhold or withdraw life support
* Patient under guardianship
* Patient deprived of liberties
* Patient included in another interventional research study under consent
* Patient already enrolled in the present study in a previous episode of acute respiratory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-04-27 (Actual); Primary Completion 2021-08-10 (Actual); Study Completion 2021-08-10 (Actual)

PRIMARY OUTCOMES:
Percentage of time spent in optimal SpO2 range | 4 hours
  The optimal SpO2 range will be defined according to the SpO2 targets determined by the clinician.

SECONDARY OUTCOMES:
Percentage of time spent in sub-optimal SpO2 range | 4 hours
  SpO2 values outside the optimal range but still within an acceptable limit (2-3 percent above and below the optimal range)
Percentage of time spent out of range | 4 hours
  Above or below the suboptimal limits specified at the begginning of the study
Percentage of time with SpO2 signal available | 4 hours
  Time with SpO2 signal available
Mean SpO2/FiO2 | 4 hours
  Mean oxygenation value
ROX index | 4 hours
  Is a predictor of HFNT success/failure defined as (SpO2/FiO2)/respiratory rate
Percentage of time with SpO2 below 88 and 85 percent | 4 hours
  Duration of time with SpO2 <85 percent and <88 percent, respectively
Number of events with SpO2 below 88 and 85 percent | 4 hours
  Frequency of SpO2 decreases <85 percent and <88 percent, respectively
Mean FiO2 | 4 hours
  Mean fraction of inspired oxygen
Percentage of time with FiO2 below 40 percent and above 60% | 4 hours
  Percentage of time that FiO2 is <40 percent and >60 percent, respectively
Number of manual adjustments | 4 hours
  Frequency of manual adjustments of FiO2
Number of alarms | 4 hours
  Frequency of alarms
Patient comfort | 4 hours
  Comfort score by visual analogic scale (from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] L'Her E, Dias P, Gouillou M, Riou A, Souquiere L, Paleiron N, Archambault P, Bouchard PA, Lellouche F. Automatic versus manual oxygen administration in the emergency department. Eur Respir J. 2017 Jul 20;50(1):1602552. doi: 10.1183/13993003.02552-2016. Print 2017 Jul. PMID 28729473
- [Background] Helmerhorst HJ, Roos-Blom MJ, van Westerloo DJ, de Jonge E. Association Between Arterial Hyperoxia and Outcome in Subsets of Critical Illness: A Systematic Review, Meta-Analysis, and Meta-Regression of Cohort Studies. Crit Care Med. 2015 Jul;43(7):1508-19. doi: 10.1097/CCM.0000000000000998. PMID 25855899
- [Background] Arnal JM, Garnero A, Novotni D, Corno G, Donati SY, Demory D, Quintana G, Ducros L, Laubscher T, Durand-Gasselin J. Closed loop ventilation mode in Intensive Care Unit: a randomized controlled clinical trial comparing the numbers of manual ventilator setting changes. Minerva Anestesiol. 2018 Jan;84(1):58-67. doi: 10.23736/S0375-9393.17.11963-2. Epub 2017 Jul 5. PMID 28679200
- [Derived] Roca O, Caritg O, Santafe M, Ramos FJ, Pacheco A, Garcia-de-Acilu M, Ferrer R, Schultz MJ, Ricard JD. Closed-loop oxygen control improves oxygen therapy in acute hypoxemic respiratory failure patients under high flow nasal oxygen: a randomized cross-over study (the HILOOP study). Crit Care. 2022 Apr 14;26(1):108. doi: 10.1186/s13054-022-03970-w. PMID 35422002